CLINICAL TRIAL: NCT06432478
Title: Study of 3D-printed Custom Applicators for Intracavitary HDR Gynaecological Brachytherapy (DISCO)
Brief Title: 3D Printed Custom Applicators for HDR BT (DISCO)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal North Shore Hospital (Other)
Collaborators: Northern Sydney and Central Coast Area Health Service (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DISCO
Record Dates: First submitted 2024-01-11; First posted 2024-05-29 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Gynecologic Cancer; Endometrial Cancer; Vaginal Cancer; Vulva Cancer
Keywords: 3D-printed applicator; Gynaecological Cancer; Brachytherapy
MeSH Terms: conditions — Endometrial Neoplasms; Vaginal Neoplasms; Vulvar Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gynaecological HDR brachytherapy patients (Experimental): Using 3D-printed custom applicators to treat gynaecological HDR brachytherapy patients
  Interventions: Device: 3D-printed custom applicator

INTERVENTIONS:
Device: 3D-printed custom applicator — 3D-printed custom applicator

SUMMARY:
Intracavitary brachytherapy for gynaecological cancer currently use cylinder-type applicators or custom wax moulds to place a radioactive source in close proximity to the treatment area and provide highly conformal dose distributions. This study is a Phase IIa non-randomised interventional pilot trial that will investigate the feasibility of successfully treating patients with 3D-printed custom applicators.

DETAILED DESCRIPTION:
Intracavitary brachytherapy for gynaecological cancer currently use cylinder-type applicators or custom wax moulds to place a radioactive source in close proximity to the treatment area and provide highly conformal dose distributions. Current workflows for designing and constructing custom applicators with wax moulds are complex, time consuming and can result in a device that fails to meet original design specifications dictated by the planning system. In contrast, 3D-printed custom applicators provide the ability to design and print patient-specific devices that match optimal design specifications. The workflow for 3D-printed applicators is also more efficient with lower turn-around time and labour/equipment costs, and ensures a more robust product for treatment. Despite these advantages there is currently no radiotherapy department offering 3D printed custom applicators at present. This study will investigate the feasibility of successfully treating gynaecological cancers with 3D-printed custom applicators.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent
* Patients indicated for intracavitary brachytherapy
* FIGO stage I-IVA
* ECOG 0-2
* Primary endometrial cancer, primary vaginal cancer, primary vulva cancer, recurrent gynaecological cancer

Exclusion Criteria:

* Pregnancy
* Patients contraindicated for brachytherapy
* Inflammatory bowel disease/history of adhesions/bowel obstruction
* Renal transplant/horseshoe kidney
* Patients with significant LVSI or pelvic sidewall invasion
* Patients requiring interstitial brachytherapy implants

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-11-24 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Successful treatment of gynaecological HDR brachytherapy patients with 3D printed intracavitary applicators. | 5 years
  To demonstrate the feasibility of successfully simulating, planning and treating a HDR BT gynaecological patient with a 3D-printed internal mould, such that there is a dosimetric and/or clinical benefit for the patient relative to the current standard of care (cylindrical vaginal applicator). Successful treatment indicated by achieving no adverse events or difference to standard of care, and dosimentic comparisons of the 3D printed applicator plan to the cylinder plan are equivalent or better. Feasibility also determined by achieving no logistical or design issues in using the 3D printed applicators clinically.

SECONDARY OUTCOMES:
To assess the patients radiation therapy acute and late toxicities using the CTCAE criteria | 5 years
  RT acute and late side effects will be assessed and quantified using CTCAE criteria via clinician assessment and PROs
To compare quality of treatment plans generated for 3D-printed moulds and cylindrical applicators assessed by dosimetric indices, statistical analysis (p-value) and comparison with international guidelines. | 5 years
  The plan quality of treatment plans generated for 3D-printed moulds and cylindrical applicators will be compared using dosimetric indices including target coverage (D90, Dose Homogeneity index) and organs at risk doses (D2cc, D1cc and point max) as well as patient comfort. statistical analysis (p-value) and comparison with international guidelines will be used to assess the quality of the treatment plans.
Determine feasibility of a pre-planned MR-only procedure | 5 years
  Feasibility of a pre-planned MR-only procedure will be determined using any of the patients that are accrued to the study who have both a CT and MRI performed at the time of simulation. The applicator and treatment plan will be generated based on the MRI and both compared to the CT-based plan and applicator. Feasibility will be indicated by generating equivalent plan quality and applicators from both methods.
To determine the feasibility of an initial CT-only process by comparing initial and final CT plan dosimetry assessed by dosimetric indices, clinical tolerances, and statistical analysis (p-value). | 5 years
  The initial and final CT plan dosimetry will be compared to determine the feasibility of an initial CT-only process. Clinically insignificant differences between the plan dosimetry metrics and all within clinical tolerances will be used to quantify the difference. statistical analysis (p-value) will be used to assess the quality of the treatment plans.
Determine feasibility of optimising 3D-printed applicator design based on the cylinder fitting procedure | 5 years
  The feasibility of an optimised 3D-printed applicator design based on the cylinder fitting procedure will be assessed by comparison of the 3D-printed clinical applicators with applicators derived from CT/MR of the vault in a relaxed state with an expansion applied based on the size of the cylinder applied in the fitting procedure. Feasibility will be determined by looking for a correlation between the size of the 3D printed clinical applicators and the size of the cylinders tolerated by the patient in the fitting procedure.
To measure resources such as procedure times and demonstrate acceptable timescales for the process | 5 years
  Procedure times will be recorded as per ARIA carepath tasks and time taken within the 3D-printed custom applicator workflow compared to the standard of care cylinder applicator workflow with equivalent or less time taken deemed acceptable
To define the resource costs associated with the 3D-printed design process and perform a cost comparison with the standard of care process | 5 years
  Costs associated with the 3D-printed design process will be defined and compared with the standard of care process via economic analysis of the resourcing and unit-price estimates in each arm of the respective workflows
To assess patient experience and acceptability of the process with questionnaires | 5 years
  Patient experience and acceptability of the 3D-printed simulation and treatment processes will be assessed with the EORTC QLQ-C30 questionnaires and success measured by comparison with the standard of care vaginal cylinder process. Questionnaires include questions with a scale of 1-4 where a higher number indicates a worse experience and a scale of 1-7 where a lower number indicates a worse experience.

CONTACTS AND LOCATIONS:
Overall Officials: Marita Morgia, MD, Principal Investigator — Royal North Shore Hospital; Jeremy Booth, PhD QMP, Study Director — Royal North Shore Hospital
Locations (1):
- Royal North Shore Hospital, St Leonards, New South Wales, Australia